CLINICAL TRIAL: NCT01213160
Title: A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of AZD4547 in Japanese Patients With Advanced Solid Malignancies
Brief Title: Study to Assess Safety and Tolerability of AZD4547 in Japanese Patient
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: D2610C00002
Record Dates: First submitted 2010-09-30; First posted 2010-10-01 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Cancer; Advanced Solid Malignancies
Keywords: Phase I; cancer; solid tumours; advanced solid malignancies; dose escalation; FGFR TKI; Japanese
MeSH Terms: conditions — Neoplasms | interventions — AZD4547

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- AZD4547 (Experimental)
  Interventions: Drug: AZD4547

INTERVENTIONS:
Drug: AZD4547 — film coated tablet, PO, twice daily

SUMMARY:
The primary purpose of this study is to explore the safety and tolerability of AZD4547 in Japanese patients with advanced solid malignancies.

DETAILED DESCRIPTION:
A Phase I, Open-Label, Multicentre Study to Assess the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-tumour Activity of Ascending Doses of AZD4547 in Japanese Patients with Advanced Solid Malignancies.

ELIGIBILITY:
Inclusion Criteria:

- Japanese patients with advanced solid malignancies Over 25 years old Relatively good overall health other than cancer

Exclusion Criteria:

- Poor bone marrow function (not producing enough blood cells). Poor liver or kidney function. Refractory nausea and vomiting, chronic gastrointestinal diseases, inability to swallow the IP or previous significant bowel resection.

Ages: 25 Years to 150 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2010-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Assessment of adverse events (based on Common Terminology Criteria for Adverse Events (CTCAE) version 4.0)general examination | General examination prior to IP administration in treatment cycles
Assessment of adverse events (based on CTCAE version 4.0)general examination | General examination on day 1 in cycle 0
Assessment of adverse events (based on CTCAE version 4.0)general examination | General examination day 21 in cycle 1.
Assessment of adverse events (based on CTCAE version 4.0), laboratory values | Laboratory assessment prior to IP administration in all treatment cycles
Assessment of adverse events (based on CTCAE version 4.0), laboratory values | Laboratory assessment on day 1 in cycle 0
Assessment of adverse events (based on CTCAE version 4.0), laboratory values | Laboratory assessment day 1 cycle 1.
Assessment of adverse events (based on CTCAE version 4.0), laboratory values | Laboratory assessment day 8 cycle 1.
Assessment of adverse events (based on CTCAE version 4.0), laboratory values | Laboratory assessment day 15 cycle 1.
Assessment of adverse events (based on CTCAE version 4.0), laboratory values | Laboratory assessment day 21 cycle 1.
Assessment of adverse events (based on CTCAE version 4.0), vital sign measurements | Vital sign measurements prior to IP administration in all treatment cycles
Assessment of adverse events (based on CTCAE version 4.0), vital sign measurements | Vital sign measurements day 1 in cycle 0
Assessment of adverse events (based on CTCAE version 4.0), vital sign measurements | Vital sign measurements day 2 in cycle 0
Assessment of adverse events (based on CTCAE version 4.0), vital sign measurements | Vital sign measurements day 8 in cycle 1.
Assessment of adverse events (based on CTCAE version 4.0), vital sign measurements | Vital sign measurements day 21 in cycle 1.
Assessment of adverse events (based on CTCAE version 4.0), left ventricular ejection fraction (LVEF) | LVEF prior to study administration
Assessment of adverse events (based on CTCAE version 4.0), LVEF | LVEF on day 21 in cycle 1.
Assessment of adverse events (based on CTCAE version 4.0), eye examination | Eye examination prior to study administration
Assessment of adverse events (based on CTCAE version 4.0), eye examination | Eye examination on day 21 in cycle 1.

SECONDARY OUTCOMES:
Define the maximum tolerated dose (MTD) if possible or biological effective dose. | Up to 3 weeks
To explore the pharmacokinetics (PK) of AZD4547and metabolite in Japanese patients with advanced solid malignancies when given AZD4547 orally. | Schedule of PK assessment 1. AZD4547; blood Cycle0-day1 -day21; 27 point 2. AZD4547 metabolite; blood Cycle1-day21; 1 poin 3. AZD4547; urine Cycle1-day21; 1 point
To obtain a preliminary assessment of the anti-tumour effect of AZD4547 by evaluation of tumour response using Response Evaluation Criteria in Solid Tumours (RECIST) criteria v1.1. | Schedule of CT/MRI etc-screeing-cycle1 day21-every 6 weeks-the end of treatment

CONTACTS AND LOCATIONS:
Overall Officials: Paul Stockman, Study Director — AstraZeneca; Hideo Saka, MD, PhD, Principal Investigator — National Hospital Organisation Nagoya Medical Centre; Yasuo Takahashi, MD, Principal Investigator — National Hospital OrganisationHokkaido Cancer Centre
Locations (3):
- Japan (3):
  - Research Site, Chūōku
  - Research Site, Nagoya
  - Research Site, Sapporo

REFERENCES:
- [Derived] Saka H, Kitagawa C, Kogure Y, Takahashi Y, Fujikawa K, Sagawa T, Iwasa S, Takahashi N, Fukao T, Tchinou C, Landers D, Yamada Y. Safety, tolerability and pharmacokinetics of the fibroblast growth factor receptor inhibitor AZD4547 in Japanese patients with advanced solid tumours: a Phase I study. Invest New Drugs. 2017 Aug;35(4):451-462. doi: 10.1007/s10637-016-0416-x. Epub 2017 Jan 10. PMID 28070720
- See also: CSR Synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=1282&filename=D2610C00002_CSR_Synopsis.pdf